CLINICAL TRIAL: NCT07217561
Title: Doula Link for Perinatal Mental Health - Trial
Brief Title: Testing "Doula Link", a Multi-Component Intervention to Improve Perinatal Mental Health
Acronym: Doula Link
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elysia Larson, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BIDMC2023P000426; K01MH133966 (NIH)
Record Dates: First submitted 2025-10-03; First posted 2025-10-16 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Perinatal Depression; Perinatal Anxiety
Keywords: Doulas; Perinatal mental health; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doula Link (Experimental): Doulas randomized to this arm will receive: 1) a doula-specific mental health toolkit; 2) training to implement an evidence-based, stress-reduction program called Our Babies and Us; 3) training for, and access to expert consultations with perinatal psychiatric specialists through MCPAP for Moms; 4) training on perinatal mental health; 5) access to doula support groups
  Interventions: Behavioral: Doula Link
- Doula Support as Usual (No Intervention): Doulas randomized to this arm will continue to provide care as usual

INTERVENTIONS:
Behavioral: Doula Link — 1) a doula-specific mental health toolkit; 2) training to implement an evidence-based, stress-reduction program called Our Babies and Us; 3) training for, and access to expert consultations with perinatal psychiatric specialists through MCPAP for Moms; 4) training on perinatal mental health; 5) access to doula support groups
  Arms: Doula Link

SUMMARY:
Doulas are trained individuals who offer informational, emotional, and physical support to their pregnant, birthing, and postpartum clients. The goal of this clinical trial is to learn if a new intervention (called "Doula Link") is feasible to implement and acceptable to both doulas and their clients. The main questions it aims to answer are:

* Is Doula Link feasible to implement and acceptable to doulas and their clients?
* What are the preliminary differences in depression and anxiety between individuals working with doulas who received Doula Link compared to those who did not receive Doula Link?

Researchers will compare "Doula Link" to usual doula practice to see if Doula Link is feasible and has potential to improve mental health outcomes in postpartum individuals.

Doulas will be randomly assigned to either receive "Doula Link" or continue with their practice as usual.

Participating doulas assigned to Doula Link will receive training mental health and implementing an intervention called "Our Babies and Us"; receive access to a toolkit; receive access to perinatal psychiatrists and referral specialists for consultations; receive access to a support group

All participating doulas will be invited to complete surveys about their experience with Doula Link (if assigned to that group) and their experience providing care for their clients.

All participating clients (pregnant and postpartum individuals) will be invited to complete surveys about their experiences with their doulas, their own mental health, and their experiences with the health system.

DETAILED DESCRIPTION:
Many people experience anxiety, depression, or other mental health concerns during the pregnancy, birth, and the postpartum periods. Despite interventions that work to prevent and treat, most perinatal depression and anxiety is unprevented and untreated. Doulas are trained professionals who offer emotional, educational, and physical support during this period. Their support has been shown to improve health outcomes for pregnant and postpartum individuals.

This study will pilot test a multi-component intervention, called Doula Link for Perinatal Mental Health (Doula Link), that gives doulas the tools to directly support mental health. Through Doula Link, doulas will receive:

1. a doula-specific mental health toolkit adapted from MCPAP for Moms, a statewide psychiatry access program;
2. training to implement an evidence-based, stress-reduction program called Our Babies and Us;
3. access to expert consultations and client referrals with perinatal psychiatric specialists through MCPAP for Moms.
4. training on perinatal mental health
5. access to doula support groups

By bringing together clinicians, doulas, and families, the goal of Doula Link is to support doulas to support their clients' mental health. Investigators hypothesize that building a program with doulas to provide direct support and link health system and community resources is an attainable intervention to expand access to mental health support.

ELIGIBILITY:
Inclusion Criteria:

* For doulas: currently providing prenatal or postpartum support to at least one client; plant to provide prenatal or postpartum support to at least three clients in the next six months; work in Massachusetts; did not participate in development of the intervention; available to participate in in-person training; English language fluency
* For clients: Pregnant or no more than 12 weeks postpartum at enrollment; served by one of the 30 study doulas; live in, and plan to give birth in Massachusetts; fluency in either English or Spanish

Exclusion Criteria:

* Not meeting inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure | 32-weeks gestation and 6 weeks postpartum postpartum for clients. Directly following, 6-months after, and 12-months after training for doulas.
  Perception among postpartum individuals in the Doula Link arm that Doula Link is agreeable and perception among postpartum individuals in the Doula Link arm that Doula Link and its individual components is agreeable. The "Acceptability of Intervention Measure (AIM) will be used. This is a four-question scale scored on a range from 1-5 with higher values indicating better acceptability.
Feasibility of Intervention | Directly following, 6-months after, and 12-months after doula training
  How well Doula Link and its individual components can be successfully delivered to doulas.
  The "Feasibility of Intervention Measure" (FIM) will be used. This is a four-question scale scored on a range from 1-5 with higher values indicating better feasibility.

SECONDARY OUTCOMES:
Appropriateness of Intervention | 32-weeks gestation and 6 weeks postpartum for clients. Directly following, 6-months after, and 12-months after training for doulas.
  The perceived fit and relevance of Doula Link and its individual components among doulas and their clients in the Doula Link arm.
  The "Appropriateness of Intervention Measure" (IAM) will be used. This is a four-question scale scored on a range from 1-5 with higher values indicating better appropriateness.
Fidelity of implementation of Our Babies and Us | Every two weeks after client enrollment for a total of six time points.
  The degree to which the Our Babies and Us component of Doula Link is implemented by the doulas to each client. This will be measured using the Our Babies and Us fidelity scale, which measures each topic across three dimensions. Possible scores range from 0 to 6 with higher scores indicating higher fidelity.
Reach of Our Babies and Us component | At 6 weeks postpartum
  The proportion of clients who receive part or all of the Our Babies and Us component of the intervention.
Symptoms of depression | 32-weeks gestation, 6-weeks postpartum, and 16-weeks postpartum
  Client scores on the Edinburgh Postnatal Depression Scale (EPDS). Possible range of scores is 0 to 30 with higher scores indicating a worse outcome.
Symptoms of anxiety | 32-weeks gestation and 6- and 16-weeks postpartum
  Symptoms of anxiety as measured by the generalized anxiety scale (GAD-7). The possible range of scores is 0 to 21 with higher scores indicating a worse outcome.
Feasibility of Our Babies and Us | Directly following, 6-months after, and 12-months after doula training
  How well doulas can implement the our Babies and Us component to their clients. The "Feasibility of Intervention Measure" (FIM) will be used. This is a four-question scale scored on a range from 1-5 with higher values indicating better feasibility.
Reach of MCPAP for Moms component | At the completion of the doula intervention
  The proportion of doulas who call to access the MCPAP for Moms component of the intervention.

OTHER OUTCOMES:
Help-seeking | 32-weeks gestation and 6- and 16-weeks postpartum
  Clients scores on the barriers to access to care evaluation scale (BACE). The possible range of scores on the BACE is 0 to 90 with higher scores indicating a worse outcome, i.e. more barriers to access to care.
Treatment participation | 32-weeks gestation and 6- and 16-weeks postpartum
  Proportion of individuals who have symptoms of depression (denominator) who report accessing treatment (numerator) in the past six weeks.
  Denominator is defined as a score of 10 or higher on the Edinburgh Postpartum Depression Scale (EPDS), indicating any thoughts of self-harm on the EPDS, or having been diagnosed with depression by a clinician.
  Numerator is defined as having seen a mental health professional or been prescribed medication to treat a perinatal mental health disorder.
Skills used | 32-weeks gestation, 6-weeks postpartum, and 16-weeks postpartum
  Our babies and us stress reduction skill used. The "Mothers and Babies Skills Utilization Scale" will be used. This 11-item scale assesses aspects of skills using a five-point frequency Likert scale. The full scale has a possible range of 0 to 44 with higher scores indicating a better outcome, i.e. more skills used.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Per institutional policy, IPD cannot be shared with other researchers without a formal data use agreement.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Larson E. Cornely RM, Gebel C, Falade E, Ezekwesili C, Peprah-Wilson S, Dodge LE, Julce C, Byatt N. A qualitative study of doulas providing emotional support during the perinatal period: an unharnessed opportunity in the United States. SSM-Health Systems 2025;4. doi: 10.1016/j.ssmhs.2025.100077
- [Background] Bohren MA, Hofmeyr GJ, Sakala C, Fukuzawa RK, Cuthbert A. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2017 Jul 6;7(7):CD003766. doi: 10.1002/14651858.CD003766.pub6. PMID 28681500
- [Background] Byatt N, Biebel K, Moore Simas TA, Sarvet B, Ravech M, Allison J, Straus J. Improving perinatal depression care: the Massachusetts Child Psychiatry Access Project for Moms. Gen Hosp Psychiatry. 2016 May-Jun;40:12-7. doi: 10.1016/j.genhosppsych.2016.03.002. Epub 2016 Mar 21. PMID 27079616
- [Background] Tandon SD, Ward EA, Hamil JL, Jimenez C, Carter M. Perinatal depression prevention through home visitation: a cluster randomized trial of mothers and babies 1-on-1. J Behav Med. 2018 Oct;41(5):641-652. doi: 10.1007/s10865-018-9934-7. Epub 2018 May 15. PMID 29766470
- [Background] Singla DR, Lawson A, Kohrt BA, Jung JW, Meng Z, Ratjen C, Zahedi N, Dennis CL, Patel V. Implementation and Effectiveness of Nonspecialist-Delivered Interventions for Perinatal Mental Health in High-Income Countries: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 May 1;78(5):498-509. doi: 10.1001/jamapsychiatry.2020.4556. PMID 33533904
- [Background] Dennis CL, Chung-Lee L. Postpartum depression help-seeking barriers and maternal treatment preferences: a qualitative systematic review. Birth. 2006 Dec;33(4):323-31. doi: 10.1111/j.1523-536X.2006.00130.x. PMID 17150072
- [Background] Byatt N, Xiao RS, Dinh KH, Waring ME. Mental health care use in relation to depressive symptoms among pregnant women in the USA. Arch Womens Ment Health. 2016 Feb;19(1):187-91. doi: 10.1007/s00737-015-0524-1. Epub 2015 Apr 7. PMID 25846018
- [Background] O'Connor E, Senger CA, Henninger ML, Coppola E, Gaynes BN. Interventions to Prevent Perinatal Depression: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2019 Feb 12;321(6):588-601. doi: 10.1001/jama.2018.20865. PMID 30747970
- [Background] Dennis CL, Falah-Hassani K, Shiri R. Prevalence of antenatal and postnatal anxiety: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):315-323. doi: 10.1192/bjp.bp.116.187179. Epub 2017 Mar 16. PMID 28302701
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562